CLINICAL TRIAL: NCT04505865
Title: The Effect of Mindfulness on Vascular Inflammation in Stable Coronary Disease: A Multi-System PET/MRI Study
Brief Title: The Effect of Mindfulness on Vascular Inflammation in Stable Coronary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael T. Osborne, Instructor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020A002750
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Atherosclerosis; Stress; Inflammation
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Optimally tolerated medical therapy
- Stress reduction (Experimental): Optimally tolerated medical therapy and stress reduction course for 8 weeks
  Interventions: Behavioral: Stress Reduction

INTERVENTIONS:
Behavioral: Stress Reduction — The stress reduction program is a multimodal mind-body resiliency program that incorporates 3 core components into each session:
  1) Elicitation of the Relaxation Response through mind-body techniques; 2) discussion about stress awareness to learn how to identify personal stressors and experiences of stress; and 3) coping strategies and adaptive perspective-taking to promote positive well-being.
  Other Names: SMART-3RP
  Arms: Stress reduction

SUMMARY:
This study aims to evaluate the effect of 8 weeks of a stress reduction intervention on atherosclerotic plaque inflammation in adults with stable coronary artery disease, as quantified by positron emission tomography (PET) with 18F-fluorodeoxyglucose (FDG) in individuals with increased psychosocial stress.

DETAILED DESCRIPTION:
This randomized controlled imaging study will be performed to evaluate the impact of mindfulness-based stress reduction via a mind body program on arterial inflammation in individuals with self-identified high levels of stress and stable coronary artery disease. Individuals will undergo baseline FDG-PET and magnetic resonance imaging (MRI) and will then be randomized to the stress-reduction intervention group or no intervention groups by blocks (1:1) with stratification by age and sex. The stress reduction sessions focus on developing an understanding of stress physiology and the physiology of the relaxation response, on developing a regular practice of eliciting the relaxation response, and on learning cognitive behavioral and positive psychology/resilience skills.

During the screening period, patient acceptability for the study will be assessed based on medical history, concomitant medications, physical examination, and clinical laboratory test results. Acceptability for study participation will be confirmed for subjects who identify as having increased levels of stress and/or a Perceived Stress Scale (PSS) score >=14. Once the patient has passed screening, they will undergo baseline imaging followed by randomization and group assignment. Approximately 12 weeks after randomization, all individuals will return for follow-up imaging and evaluation.

FDG PET/MRI scans will be performed during the study for baseline and follow up to assess the intervention's impact on the brain as well as systemic and arterial inflammation along with other changes in related biomarker and imaging parameters. The Perceived Stress Scale will be delivered prior imaging during both imaging visits to measure perceived psychological stress. During both imaging sessions, subjects will be exposed to overt faces to measure signals during brain imaging.

ELIGIBILITY:
Inclusion Criteria:

* Must admit to feeling stressed and/or have PSS score > 13 (moderate stress)
* Must be willing to complete stress reduction course and imaging sessions with < 3 missed appointments in last year
* Known clinical cardiovascular disease with prior atherosclerotic myocardial infarction, percutaneous intervention or bypass surgery > 6 months before entry, or severe coronary calcifications on computed tomography or coronary calcium score >400
* Stable symptoms without symptomatic heart failure or arrhythmia or planned revascularization
* Maximally tolerated and stable medical regimen for 90 days that does not include a high intensity statin for clinical reasons
* No neurological disease or systemic inflammatory disease/current anti-inflammatory therapy
* No active psychiatric disease/medications or substance abuse (including tobacco smoking or more than moderate alcohol) for last 6 months
* No current participation in cardiac rehab or prior participation in stress reduction
* For imaging: no pregnancy, weight > 300 lbs., metal implants, uncontrolled hyperglycemia, or inability to provide consent or comply

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in arterial inflammation by PET imaging | 12 weeks
  Change in arterial inflammation measured as the ratio of tracer activity in the walls of the aorta and carotid arteries to the activity of background venous blood on FDG PET imaging (ratio without units) - from initial imaging to repeat imaging

SECONDARY OUTCOMES:
Change in brain activity by PET | 12 weeks
  Change in brain activity ratio of tracer activity in the amygdala (a stress-associated brain center) to the activity of background brain cortical tissue on FDG PET imaging (ratio without units) based on FDG PET - from initial imaging to repeat imaging
Change in bone marrow activity by PET | 12 weeks
  Change in bone marrow activity measured in the vertebral bodies as a mean standardized uptake value (g/mL) based on FDG PET - from initial imaging to repeat imaging
Change in inflammatory biomarkers | 12 weeks
  Change in high-sensitivity C-reactive protein (mg/L)- from initial imaging to repeat imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Osborne, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes